CLINICAL TRIAL: NCT06173622
Title: Effects of Fetal Positioning on Pain and Physiological Parameters During Venipuncture in Preterm Neonates: A Randomized Controlled Trial
Brief Title: Effects of Fetal Positioning During Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Evrim Kızıler, Assistant Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EKIZILER-001
Record Dates: First submitted 2023-11-25; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Preterm Neonates; Venipuncture
Keywords: Preterm neonates; Venipuncture; Fetal positioning; Pain; Physiological parameters; Nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fetal positioning group (Experimental): The neonates in the experimental group were put into fetal positioning at least 10 minutes before the procedure, and then venipuncture was performed. The fetal positioning was maintained throughout the procedure and the patient was kept in the fetal position for at least five more minutes after needle removal.
  Interventions: Behavioral: Fetal Positioning
- Control group (No Intervention): No intervention was performed by the researchers on the neonates included in the control group, and venipuncture was performed in accordance with the standard procedure of the neonatal intensive care unit.

INTERVENTIONS:
Behavioral: Fetal Positioning — In the study, venipuncture was applied to the intervention and control groups. While the procedure was performed by an experienced neonatal nurse, the neonates' pain score, crying duration and physiological parameters were monitored by another researcher (observer).
  Arms: Fetal positioning group

SUMMARY:
The study was aimed to examine the effects of fetal positioning during venipuncture on the neonates' pain score and physiological parameters (heart rate, blood-oxygen saturation, body temperature, crying duration) in neonatal intensive care unit (NICU).

This randomized controlled clinical trial was conducted between 10.2021-07.2022 with 60 preterm neonates, aged 26-32 week of gestation. Neonates were divided into intervention group (n=30) and control group (n=30) according to the randomization method. The neonates in the intervention group were put into fetal positioning at least 10 minutes before the procedure, and then venipuncture was performed. The fetal positioning was maintained throughout the procedure and the patient was kept in the fetal position for at least five more minutes after the procedure. Changes in the neonates' pain score and crying duration as well as heart rate, blood temperature, blood-oxygen saturation at three time points: before the procedure, immediately after needle insertion, five minutes after needle removal. Data was collected using the sociodemographic form, neonatal observation form and Neonatal Pain, Agitation and Sedation Scale (N-PASS). The collected data were analyzed using the SPSS 15 software.

The main questions it aims to answer:

1. Does fetal positioning have an effect on pain score of premature neonates?
2. Does fetal positioning have an effect on heart rate of preterm neonates?
3. Does fetal positioning have an effect on oxygen saturation of preterm neonates?
4. Does fetal positioning have an effect on body temperature of the preterm neonates?
5. Does fetal positioning have an effect on the crying duration of preterm neonates?

DETAILED DESCRIPTION:
Neonates who were hypotonic, lethargic, in shock or had seizures, stage 3-4 intracranial hemorrhage and a history of surgery were not included in the study. Additionally, neonates was taken any analgesic and/or sedative in the last 24 hours were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns (a) whose parents volunteered to participate in the study, (b) required venipuncture, and (c) were born at 26-32 gestational weeks were included in the study.

Exclusion Criteria:

* Newborns who are hypotonic, lethargic, in shock or having seizures,
* Newborns with a history of stage 3-4 intracranial hemorrhage
* Newborns with a history of surgery
* Newborns whose gestational week is over 37 weeks
* Newborns who have taken any analgesics and/or sedatives in the last 24 hours,
* Newborns who have had any invasive procedure within the last hour
* Newborns whose parents do not volunteer

Ages: 6 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Pain score | Before the procedure, immediately after needle insertion, five minutes after needle removal.
  Neonatal Pain Agitation and Sedation Scale (N-PASS) is a multidimensional scale that scores 5 behavioral and physiologic parameters for both pain and sedation. It is proficient in assessing continuous, acute, and chronic pain. In the scale crying/irritability, behavior state, facial expression, ekstremites tone and vital signs of newborns are scored between 0-2 points and the total score is obtained. A minimum of 0 and a maximum of 10 points are obtained from the scale, and an increase in score indicates an increase in pain. A score of four and below reflects mild pain, and a score of five and above reflects moderate and severe pain.
Heart rate | Before the procedure, immediately after needle insertion, five minutes after needle removal.
  The newborn's heart rate was monitored with a neonatal monitor and recorded on the monitoring form.
Oxygen saturation | Before the procedure, immediately after needle insertion, five minutes after needle removal.
  The neonates' oxygen saturation was monitored with a neonatal monitor and recorded on the monitoring form.
Body temperature | Before the procedure, immediately after needle insertion, five minutes after needle removal.
  The neonates' body temperature was monitored with a neonatal monitor and recorded on the monitoring form.

SECONDARY OUTCOMES:
Crying duration | Before the procedure, immediately after needle insertion, five minutes after needle removal.
  The newborn's crying duration was recorded by the researcher (observer) using a chronometer.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim KIZILER, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Evrim KIZILER, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez O, Subramanian P, Rahmat N, Theam LC, Chinna K, Rosli R. The effect of facilitated tucking on procedural pain control among premature babies. J Clin Nurs. 2015 Jan;24(1-2):183-91. doi: 10.1111/jocn.12657. Epub 2014 Jul 24. PMID 25060423
- [Result] Holsti L, Grunau RE, Whifield MF, Oberlander TF, Lindh V. Behavioral responses to pain are heightened after clustered care in preterm infants born between 30 and 32 weeks gestational age. Clin J Pain. 2006 Nov-Dec;22(9):757-64. doi: 10.1097/01.ajp.0000210921.10912.47. PMID 17057556
- [Result] Liaw JJ, Yang L, Katherine Wang KW, Chen CM, Chang YC, Yin T. Non-nutritive sucking and facilitated tucking relieve preterm infant pain during heel-stick procedures: a prospective, randomised controlled crossover trial. Int J Nurs Stud. 2012 Mar;49(3):300-9. doi: 10.1016/j.ijnurstu.2011.09.017. Epub 2011 Oct 14. PMID 22001561